CLINICAL TRIAL: NCT00138255
Title: MMR and Varicella Vaccine Responses in Extremely Premature Infants
Brief Title: Responses of Premature Infants to Measles-Mumps-Rubella (MMR) and Varicella Vaccines
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 03-140
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-05

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to see if the MMR and chickenpox vaccines work as well in premature infants as in children that were carried to full term. A group of children who were carried full-term will be matched for age, sex, and race and will be used for comparison.

DETAILED DESCRIPTION:
The purpose of this study is to see if the MMR and chickenpox vaccines work as well in premature infants as in children that were carried to full term. A group of children who were carried full-term will be matched for age, sex, and race and will be used for comparison. Extremely premature infants (born at <28-30 weeks gestation) have lower antibody responses than full-term infants to several vaccines given at the postnatal ages recommended for full term infants. We propose to evaluate the immunogenicity of varicella and mumps-measles-rubella (MMR) vaccines in relatively healthy 15 month-old children born at <29 weeks gestation. This is a phase IV, observational study with 2 study arms having 16 infants each. The first group will enroll infants 9-12 months old that were born premature (<29 weeks gestation). The second group will be matched for sex, race, and postnatal age, but will have been full term (>= 37 weeks gestation) at birth. Infants will be vaccinated at visit 1 and post-vaccine serology will drawn at visit 2 (4 to 6 weeks after visit 1).

ELIGIBILITY:
Inclusion Criteria:

1. Premature infant < 29 weeks gestation at birth or term infant >= 37 weeks gestation at birth.
2. Postnatal age < 16 months, 0 days.
3. Has not yet received MMR or varicella vaccines. (There are no restrictions on the administration of other vaccines at the time of MMR/varicella vaccination.)
4. Parental permission.
5. Agreement of primary care pediatrician/ health care provider.
6. Receives primary pediatric care within an approximate 25-mile radius of the University of Rochester.
7. Healthy status at enrollment.

Exclusion Criteria:

1. Known immunodeficiency.
2. Systemic corticosteroid therapy at the time of MMR/varicella vaccination.
3. Requiring oxygen therapy.
4. Clinically significant findings on review of medical history and physical exam determined by the investigator or sub-investigator to be sufficient for exclusion.
5. Any condition determined by the investigator that would interfere with the evaluation of the vaccine or be a potential health risk to the subject.

Max Age: 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32
Dates: Start 2004-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester School of Medicine and Dentistry, Rochester, New York, United States